CLINICAL TRIAL: NCT02646683
Title: An Open Label Interventional Phase 4 Study to Evaluate Efficacy, Safety and Mucosal Healing of Early Versus Late Use of Vedolizumab in Crohn's Disease: the LOVE-CD Study (LOw Countries VEdolizumab in CD Study)
Brief Title: A Study to Evaluate Efficacy, of Early Versus Late Use of Vedolizumab in Crohn's Disease: the LOVE-CD Study
Acronym: LOVE-CD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Geert D'Haens (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Geert D'Haens, Coordinating Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-100757
Record Dates: First submitted 2015-08-27; First posted 2016-01-06 (Estimated); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Crohn's disease (Other): VEDOLIZUMAB 300 mg at week 0,2,6, (10), 14, 22, 30,(34), 38, (42), 46, (50)
  week 10 = only required for subjects not responding week 34, 42 and 50- only required for subjects who have no endoscopic improvement at week 26
  Interventions: Drug: vedolizumab
- Late Crohn's disease (Other): VEDOLIZUMAB 300 mg at week 0,2,6, (10), 14, 22, 30,(34), 38, (42), 46, (50)
  week 10 = only required for subjects not responding week 34, 42 and 50- only required for subjects who have no endoscopic improvement at week 26
  Interventions: Drug: vedolizumab

INTERVENTIONS:
Drug: vedolizumab
  Other Names: Entyvio

SUMMARY:
This multi-centre open label study will involve a minimum of 260 patients in 2 cohorts: 86 patients with 'early CD' defined as disease duration < 24 months and no other treatments than corticosteroids and/or thiopurines and 174 patients with 'late CD' defined as active disease despite treatment with immunosuppressives and anti-TNF. Patients with intolerance to IS and anti-TNF will also be allowed in the latter group. Participants will be treated with 12 months of open label vedolizumab (study medication followed by commercial medication once reimbursement is available) and undergo monitoring of endoscopic, histological and clinical disease parameters. No randomization or blinding will be performed but the study management will ensure that recruitment in either study group is comparable for number and profile of patients (on/off steroids).

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic inflammatory disease of the small bowel and colon. Symptoms commonly include bloody diarrhea, abdominal pain, weight loss, and fever. There is no known cause or cure for CD. The aim of current CD treatments is to induce and maintain remission, to reduce the need of corticosteroids and avoid resections and fistulas.

Treatment options include systemic and/or topical corticosteroids, purine analogues (6-mercaptopurine and azathioprine), anti-TNF antibodies and surgery. In 2013, results from the GEMINI II, phase 3, randomized controlled trial demonstrated the efficacy of vedolizumab (VDZ) in inducing and maintaining remission in adult patients with active CD.

VDZ (MLN0002, or MLN02), inhibits the interaction between α4β7 integrin on memory T and B cells and mucosal addressin cell adhesion molecule-1 expressed on the vascular endothelium of the gut and has been shown to be effective in both inducing and maintaining clinical remission in ulcerative colitis. The ideal positioning of vedolizumab in the therapeutic armamentarium for CD remains unknown. With other (anti-TNF) biologics, outcomes have usually been better if the treatment was started earlier in the disease course and if the patients had not been exposed to prior antibody treatments. Therefore, it appears appropriate and desirable to test the potency of vedolizumab in an earlier phase of CD.

Indeed, also with vedolizumab patients previously exposed to biologics appear to have lower success rates with vedolizumab, so a position earlier in the disease course would most likely lead to better outcomes.

This is an investigator-initiated open label study of VDZ therapy in 2 distinct populations of CD patients with active disease: 1. patients who have been diagnosed < 2 years ago and who only been exposed to aminosalicylates and corticosteroids and 2. patients who have been exposed to immunomodulators and/or anti-TNF agents in addition to steroids and aminosalicylates.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements.
2. The subject signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Age 18 to 80
4. Male or non-pregnant, non-lactating females. Females of child bearing potential must have a negative serum pregnancy test prior to randomization, and must use a hormonal (oral, implantable or injectable) or barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
5. Established diagnosis of ileal, ileocolonic or colonic Crohn's disease with histopathological confirmation available in the record of the patient.
6. Moderately to severely active CD (CDAI 220-450) with objective evidence of ulcerations visualized on endoscopy.
7. Anti-TNF discontinued for at least 4 weeks prior to baseline.

   GROUP 1 (EARLY CD):
8. Diagnosis of CD < 24 months prior to enrollment
9. Demonstrated failure to respond to topical or systemic corticosteroids or intolerance to corticosteroids or: need for > 2 courses of steroids since diagnosis or: steroid dependency at any dose since diagnosis and additionally, but not mandatory, lack of efficacy of thiopurines or intolerance to thiopurines (any duration). Patients who are using thiopurines at screening must have used them for > 3 months (last 4 weeks at stable dose).

   GROUP 2 (LATE CD)
10. Demonstrated failure to respond to at least 3 months of thiopurines or intolerance to thiopurines and: failure to respond to at least 1 anti-TNF or intolerance to anti-TNF or loss of response to at least 1 anti-TNF.

Exclusion Criteria:

1. Previous exposure to any anti-integrin antibodies including- vedolizumab ; α4β7 anti-bodies ; β7 antibodies ; anti- MADCAM-1
2. Contraindication for endoscopy.
3. History of colonic dysplasia/cancer
4. Presence of stoma
5. Received other biologics within the last 4 weeks of baseline
6. Use of 5-aminosalicylic acid (5-ASA) or corticosteroid enemas/suppositories within 2 weeks of enrollment
7. Chronic hepatitis B or C infection
8. Evidence of or treatment for C. difficile infection or other intestinal pathogen at screening within 4 weeks prior to enrollment
9. Active or latent tuberculosis
10. Conditions which in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures.
11. Received any investigational drug in the past 30 days or 5 half-lives, whichever is longer.
12. Positive progressive multifocal leukoencephalopathy ( PML) subjective symptom checklist before enrollment.
13. Subjects with known allergy or hyposensitivity to vedolizumab or its components

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with clinical and endoscopic remission at Week 26 | week 26
  Crohns disease activity index (CDAI) of 150 or lower and Simple endoscopic score for Crohn's disease (SES-CD) < 4.

SECONDARY OUTCOMES:
Proportion of patients with endoscopic response at Weeks 26 and 52 | 26 and 52 weeks
  SES-CD reduction by ≥ 50 %
Proportion of patients with 25% and 75% reduction of SES-CD at Weeks 26 and 52 | 26 and 52 weeks
  SES-CD reduction
Proportion of patients with clinical response | 52 weeks
  CDAI decrease of ≥ 70 points from baseline
Proportion of patients with clinical remission | 52 weeks
  (CDAI <=150) at all time other points
Proportion of patients with corticosteroid- free clinical remission | 52 weeks
  (CDAI <=150) at all other time points
Proportion of patients with normalized serum C-reactive protein (CRP) at all time points | 52 weeks
  CRP
Proportion of patients with no granulocytes in the biopsies at Weeks 26 and 52. | Week 26 and week 52
  No granulocytes
Proportion of patients with 25%, 50% and 75% reduction in the Geboes histology score at Weeks 26 and 52 | Week 26 and week 52
  Geboes score
Proportion of patients with sustained clinical response (response at all time points after week 10) | After week 10
  Geboes score reduction
Proportion of patients with sustained clinical remission | After week 10
  (remission at all time points after week 10)
Proportion of patients with draining fistulas | 52 weeks
  Fistula
Proportion of patients that need to be hospitalized | 52 weeks
Quality of life measured by Inflammatory Bowel Disease Questionnaire ( IBDQ) | Screening, week 10, week 26 and week 52
  Questionnaire
Work productivity Index | Screening, week 10, week 26 and week 52
  Questionnaire
Serum concentrations of vedolizumab and antibodies to vedolizumab before every infusion | 52 weeks
  through concentration
Quality of life measured by Euroqol (EQ-5D) | Screening, week 10, week 26 and week 52
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Geert D'Haens, Prof, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (23):
- Belgium (15):
  - UZ Antwerpen, Antwerp
  - Imeldahospital, Bonheiden
  - AZ Sint-Lucas, Bruges
  - ULB Erasme, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Sint Lucas, Ghent
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHC Clinique Saint-Joseph, Liège
  - CHU de Liège, Liège
  - ZNA Jan Palfijn, Merksem
  - AZ Damiaan, Ostend
  - AZ Delta Roeselare, Roeselare
  - St Vincentius, Wilrijk
- Hungary (3):
  - Semmelweis University, Budapest
  - University of Debrecen, Debrecen
  - Universtiy of Szeged, Szeged
- Netherlands (5):
  - Academisch Medisch Centrum, Amsterdam
  - Ziekenhuis Gelderse Vallei, Ede
  - OLVG, Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus MC, Rotterdam

REFERENCES:
- [Derived] Hanzel J, Dreesen E, Vermeire S, Lowenberg M, Hoentjen F, Bossuyt P, Clasquin E, Baert FJ, D'Haens GR, Mathot R. Pharmacokinetic-Pharmacodynamic Model of Vedolizumab for Targeting Endoscopic Remission in Patients With Crohn Disease: Posthoc Analysis of the LOVE-CD Study. Inflamm Bowel Dis. 2022 May 4;28(5):689-699. doi: 10.1093/ibd/izab143. PMID 34137430